CLINICAL TRIAL: NCT04132453
Title: Evaluation of Sensifree's Algorithm for Continuous Blood Pressure Measurements Based on a PPG Sensor's Signal Compared to Invasive Radial Arterial Line
Brief Title: Continuous Blood Pressure and Waveform Measurements Comparison Between Invasive Arterial Line and PPG Sensor
Status: Completed | Type: Observational
Sponsor: Sensifree Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLI-0003.04
Record Dates: First submitted 2019-10-16; First posted 2019-10-18 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2020-10

CONDITIONS: Blood Pressure Measurement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Arterial catheterization kit — Invasive monitoring of blood pressure via catheterization of the radial artery, displaying a continuous pressure waveform
Device: GE Datex-Ohmeda Finger Clip Pulse Oximeter Sensor — PPG based, fingertip mounted sensor, that measures the oxygen level (oxygen saturation) of the blood and generates a waveform
Device: NIBP Cuff (GE Healthcare) — A blood pressure cuff is used to measure blood pressure. The cuff has an inflatable rubber bladder that is typically fastened around the arm. A pressure meter indicates the cuff's pressure.

SUMMARY:
The purpose of this study is to compare blood pressure values (systolic, diastolic, mean arterial pressure) and waveform as recorded by a radial arterial line catheter to the waveform and values as calculated by the Sensifree's algorithm from a PPG sensor from a variety group of patients during elective surgeries.

DETAILED DESCRIPTION:
Before induction of anesthesia, an arterial line will be inserted to the patient radial artery using a designated short, stiff tubing kit according to catheter IFU (Instructions for Use), preferably under US guidance. Removal of air bubbles from the catheter-transducer system is mandatory prior to connecting the tubing to the catheter.

Study nurse will connect a Sensifree laptop with designated data acquisition software (Medicollector BEDSIDE) to the multi-parameter monitor communication port and start the recording of invasive blood pressure and pulse oximeter pleth (PPG sensor) per software IFU. Prior to connecting the arterial line system to the patient, a calibration (flush test) will be done and recorded. During the study, any deterioration in the waveform recorded by the intra-arterial catheter will be noted and appropriate corrective measures will be taken as soon as possible (e.g., flushing or adjusting the position of the catheter).

Preferable NIBP (Non Invasive Blood Pressure) measurement rate will be every 10 minutes, unless the medical procedure requires otherwise.

Calibration procedure will be repeated every 60 +/- 5 minutes and at the end of the surgery. Recording will take place for the duration of the surgery.

NIBP cuff will be placed over the arterial-line arm, NIBP air hose will be replaced with an air hose supplied by Sensifree and the pressure gauge in it will be connected to Sensifree laptop via analog to digital converter in order to capture the data.

Medication used during the surgery will be listed and documented in the CRF (Case Report Form) including drugs name, dose, time and method of administration.

Offline data analysis will compare the blood pressure values as calculated by the Sensifree's algorithm based on the PPG signal, to the values obtained from the arterial line. The comparison results will be measured against the accuracy performance requirements per ISO 81060-2.

ELIGIBILITY:
Inclusion Criteria:

* Signed inform consent
* Age 18-20
* Elective surgery that requires invasive BP monitoring (A-line)

Exclusion Criteria:

* Emergency surgery
* Subject has a condition that might prevent BP fluctuations
* Subject is taking medicine that might prevent BP fluctuations
* Arterial line not placed in the radial artery
* Flush test has inadequate frequency response pre-trial
* Subject's arterial line contralateral hand is not available for PPG sensor placement
* Subject has 50% or more pacemaker dependency

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective surgery involving placement of radial artery A-line for BP monitoring
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Comparison of waveforms and BP values between PPG sensor and arterial line | 3 months after last patient enrolled
  Blood pressure waveform will be acquired from the PPG while blood pressure waveform and values (systolic, diastolic, mean) will be acquired from A-line. PPG data will be analyzed by the Sensifree's algorithm and compared to the A-line measurement results according to ISO 81060-2 accuracy specifications

CONTACTS AND LOCATIONS:
Overall Officials: Inbal Dabush-Elisha, MD, Principal Investigator — Wolfson Medical Center
Locations (1):
- Wolfson Medical Center, Holon, Israel

IPD SHARING:
Plan to Share IPD: No